CLINICAL TRIAL: NCT02312869
Title: Local Assessment of Management of Burn Patients (LAMiNAR) - a Prospective Observational International Multicenter Cohort Study
Brief Title: Local Assessment of Management of Burn Patients
Acronym: LAMiNAR
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: LAMiNAR
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Burns - Multiple; Mechanical Ventilation
Keywords: Mechanical Ventilation; Burn patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — not applicable, observational study

SUMMARY:
In the general intensive care unit (ICU) population, there is strong evidence for benefit from lung-protective mechanical ventilation, including the use of low tidal volumes and adequate levels of positive end-expiratory pressure (PEEP). In burn patients it is highly uncertain whether these settings are beneficial and there are even concerns over safety of, in particular use of low tidal volumes. There is lack of international guidelines and consequently ventilation practice in burn patients may widely vary.

The primary objective is to determine ventilation practice in burn ICUs worldwide, focusing on the size of tidal volumes and the levels of PEEP used for burn patients. In addition, data on other strategies considered important in patients who receive ventilation are also collected, including data on neuromuscular blocking agents, sedatives and analgesics, and type and amount of intravenous fluids used in the period of ventilation. The secondary objective is to determine the association between tidal volume size and levels of PEEP, and duration of ventilation in burn patients.

DETAILED DESCRIPTION:
Patient population: Consecutive burn patients admitted to participating burn ICUs who receive invasive ventilation, irrespective of severity of burn injury and/or presence of inhalation trauma are eligible for participation.

Data collection: includes burn patients admitted within a period of three months. Demographic and baseline data are collected from the clinical files on the day of admission. If available, standard of care and clinical outcome parameters are collected daily until day 14, death or discharge from ICU, whatever comes first.

Sample size: The primary objective is to determine (variations in) ventilation practice in burn patients in burn ICUs. Therefore, the sample size is based on the main secondary objective, which is to determine the association between the following ventilator settings: tidal volume, PEEP, FiO2 and mode; and outcome of burn patients. The investigators calculated the sample size for a multiple regression model: a sample size of at least 300 patients is required to have a power of 0.80, a significance level of 0.05, using an estimated effect size of 0.04, while using 4 independent variables in the model.

Ethics Approval: National coordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate according to local policy. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place. The investigators expect that in most, if not every participating country, a patient informed consent is not be required.

Monitoring: Due to the observational nature of the study, a DSMB is not necessary.

Organization: National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local coordinators in each site will supervise data collection and ensure adherence to Good Clinical Practice during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Burns
* Admission to a participating burn ICU Need for invasive ventilation
* Informed consent (only if applicable in the country where data are collected)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive intubated and ventilated burn patients admitted to participating ICUs during a period of 3 months
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Ventilation parameters | Up to 14 days during mechanical ventilation
  Tidal volume size; milliliters per kilogram of predicted body weight
Ventilation parameters | Up to 14 days during mechanical ventilation
  Level of positive end-expiratory pressure (PEEP); cm H2O
Ventilation parameters | Up to 14 days during mechanical ventilation
  Fraction of oxygen in inspired air (FiO2), %
Ventilation parameters | Up to 14 days during mechanical ventilation
  Mode of ventilation; assist-control or spontaneous modes of ventilation

SECONDARY OUTCOMES:
Number of ventilator-free days and alive at day 28 | From day 1 to day 28
  Defined as the number of days, from day 1 to day 28, the patient is alive and breathes without assistance of a mechanical ventilator, if the period of unassisted breathing lasted at least 24 consecutive hours. Notably, if after successful withdrawal of mechanical ventilation the patient requires ventilation for a surgical procedure, this will not count as a 'ventilator day'. If ventilation is prolonged after surgery due to respiratory insufficiency, the day(s) ventilation is required counts as a 'ventilator day'
Other Ventilation Parameters | Up to 14 days during mechanical ventilation
  Peak and plateau pressures or maximum airway pressure
Other Ventilation Parameters | Up to 14 days during mechanical ventilation
  Respiratory rate
Other Ventilation Parameters | Up to 14 days during mechanical ventilation
  Inspiration to expiration ratio
Other Ventilation Parameters | Up to 14 days during mechanical ventilation
  Peripheral oxygen saturation
Other Ventilation Parameters | Up to 14 days during mechanical ventilation
  Arterial blood gas parameters
Length of Stay in ICU on Day 90 | Until day 90
  Time between admission and discharge or death
Length of Stay in Hospital on Day 90 | Until day 90
  Time between admission and discharge or death
All-cause ICU Mortality | Until day 90
  Any death during ICU stay
All-cause Hospital Mortality | Until day 90
  Any death during hospital stay
Need for Tracheostomy | daily up to 14 days from inclusion
  Need for tracheostomy, first tracheostomy will be assessed up to 14 days from inclusion
Daily Lung Injury Scores | Up to 14 days during mechanical ventilation
  Score based on chest X-ray findings (if obtained), PaO2/FiO2, PEEP level and respiratory compliance.
Daily Sequential Organ Failure Assessment (SOFA)-scores | Daily up to 14 days from inclusion
  six-organ dysfunction/failure score measuring multiple organ failure daily
Complications | Daily up to 14 days from inclusion
  Complications will include: Skin and soft tissue infections
Complications | Daily up to 14 days from inclusion
  Complications will include: (Ventilator associated) Pneumonia
Complications | Daily up to 14 days from inclusion
  Complications will include: Sepsis
Complications | Daily up to 14 days from inclusion
  Complications will include: Acute respiratory distress syndrome according to Berlin criteria
Complications | Daily up to 14 days from inclusion
  Complications will include: Acute renal failure
Complications | Daily up to 14 days from inclusion
  Complications will include: Abdominal compartment syndrome

OTHER OUTCOMES:
Standard care strategies | Daily up to 14 days from inclusion
  Strategies considered to be important in patients who receive ventilation, including: Fluid balance, types and dose of fluids used
Standard care strategies | Daily up to 14 days from inclusion
  Strategies considered to be important in patients who receive ventilation, including: use of sedative and analgesic drugs
Standard care strategies | Daily up to 14 days from inclusion
  Strategies considered to be important in patients who receive ventilation, including: use of sedation and delirium scores
Standard care strategies | Daily up to 14 days from inclusion
  Strategies considered to be important in patients who receive ventilation, including: use of neuromuscular blocking agents
Standard care strategies | Daily up to 14 days from inclusion
  Strategies considered to be important in patients who receive ventilation, including: use of antibiotic prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J. Schultz, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Schultz MJ, Horn J, Hollmann MW, Preckel B, Glas GJ, Colpaert K, Malbrain M, Neto AS, Asehnoune K, de Abreu MG, Martin-Loeches I, Pelosi P, Sjoberg F, Binnekade JM, Cleffken B, Juffermans NP, Knape P, Loef BG, Mackie DP, Enkhbaatar P, Depetris N, Perner A, Herrero E, Cachafeiro L, Jeschke M, Lipman J, Legrand M, Horter J, Lavrentieva A, Glas G, Kazemi A, Guttormsen AB, Huss F, Kol M, Wong H, Starr T, De Crop L, de Oliveira Filho W, Manoel Silva Junior J, Grion CMC, Jeschke MG, Burnett M, Mondrup F, Ravat F, Fontaine M, Asehoune K, Floch RL, Jeanne M, Bacus M, Chaussard M, Lehnhardt M, Mikhail BD, Gille J, Sharkey A, Trommel N, Reidinga AC, Vieleers N, Tilsley A, Onarheim H, Bouza MT, Agrifoglio A, Freden F, Palmieri T, Painting LE; LAMiNAR investigators. Ventilation practices in burn patients-an international prospective observational cohort study. Burns Trauma. 2021 Dec 16;9:tkab034. doi: 10.1093/burnst/tkab034. eCollection 2021. PMID 34926707
- See also: LAMiNAR Website — https://sites.google.com/site/laminarstudy/
- See also: PROVE NETWORK Website — https://sites.google.com/site/proveneteu/provenet-studies